CLINICAL TRIAL: NCT05254782
Title: From Liquid Biopsy to Cure: Using ctDNA Detection of Minimal Residual Disease to Identify Patients for Curative Therapy After Lung Cancer Resection (ctDNALung-Detect)
Brief Title: Using ctDNA to Detect Minimal Residual Disease After Lung Cancer Resection
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Ontario Institute for Cancer Research (Other); The Princess Margaret Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 20-6199
Record Dates: First submitted 2022-02-14; First posted 2022-02-24 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue, plasma, buffy coat
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ctDNALung-Detect is an investigator-initiated single arm, multi-institution study designed to assess the ctDNA detection rate and its association with Relapse Free Survival (RFS) in operable stage T1-T4 (T3,T4 multifocal) N0M0 non-small cell lung cancer (NSCLC) patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Ability to provide written informed consent;
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
4. T1-T4 (T3,T4 multifocal) N0M0 NSCLC who are planned for complete surgical resection;
5. Tumour size must be at least 1 cm (unidimensional) and have at least some solid component on imaging;
6. Surgical tumour formalin-fixed, paraffin-embedded (FFPE) specimens for ctDNA studies are required.

Exclusion Criteria:

1. Prior radiation, surgery or chemotherapy for the current diagnosis of NSCLC is not permitted.
2. Incomplete surgical resection. Participants who had pre-operative ctDNA samples taken but subsequently do not have a complete surgical resection would not qualify for post-operative ctDNA testing.
3. Concurrent enrolment in a therapeutic study using drug or radiation therapy. Enrolment in observational, diagnostic or studies of novel surgical techniques will be allowed.
4. Concurrent active malignancy or other invasive malignancy within previous 2 years. Non-invasive malignancies (i.e., cervical carcinoma in situ, in situ prostate cancer, non-melanomatous carcinoma of the skin, ductal carcinoma in situ of the breast that has been surgically cured) are excluded from this definition.
5. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Early stage (T1-T4 (T3,T4 multifocal) N0M0) non-small cell lung cancer, with planned complete surgical resection.
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Rate of ctDNA Detection | Up to 24 Months
  The percentages of pre-operative and post-operative ctDNA detection in patients with T1-T4N0 (T3, T4 multifocal) NSCLC will be estimated together with their Clopper-Pearson exact 95% CIs.
Relapse Free Survival | Up to 36 Months
  Relapse free survival (RFS) will be estimated using the Kaplan-Meier method and compared using the logrank test among patients with and without detectable ctDNA pre- or post-operatively.

SECONDARY OUTCOMES:
Overall Survival | Up to 36 Months
  Overall survival (OS) will be estimated using the Kaplan-Meier method and compared using the log-rank test between patients with and without detectable ctDNA pre- or post-operatively.

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Michael Garron Hospital, Toronto, Ontario
  - St. Joseph's Health Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario